CLINICAL TRIAL: NCT00046696
Title: A Phase I and Pharmacokinetic Study of NM-3 Administered Orally Once or Twice Daily on Five Consecutive Days and Repeated Weekly for Six Weeks Every Eight Weeks in Patients With Advanced Solid Tumors.
Brief Title: A Study of NM-3 Administered Orally in Patients With Advanced Solid Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NM-103
Record Dates: First submitted 2002-10-01; First posted 2002-10-02 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Neoplasms
Keywords: Cancer; Cancer Alternative Therapies; Living with Cancer
MeSH Terms: conditions — Neoplasms

INTERVENTIONS:
Drug: NM-3

SUMMARY:
A study for patients who have failed standard therapy. If there is no dose limiting toxicities the patients will receive further cycles of therapy if there is no evidence of disease progression.

DETAILED DESCRIPTION:
This is a non-randomized, open-label, Phase I study. A modified Fibonacci dose escalation will be used to determine the MTD for subsequent Phase II trials. Study duration is expected to be 12 to 18 months. Patients with a histological or cytological diagnosis of a solid tumor who have failed standard therapy or for whom no standard therapy exists are enrolled. If there is no dose limiting toxicities and if patients meet the inclusion criteria and have none of the exclusion criteria of the protocol, they will receive further cycles of therapy if there is no evidence of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients at least 18 years of age.
* All patients must have an advanced solid tumor that has failed standard therapy or for which no standard therapy exists.
* Histological or cytological diagnosis of a malignant solid tumor.
* Measurable or non-measurable disease.
* Any chemotherapy, radiotherapy, or major surgery at least 4 weeks prior to study entry (6 weeks for nitrosoureas or mitomycin C). Patients must have recovered from the toxic effects of any prior therapy.
* Karnofsky performance status index greater than or equal to 80.
* Must have adequate organ and immune system function according to the study design, obtained less than or equal to 7-days prior to treatment with NM-3.
* Female patients of childbearing potential must have a negative serum pregnancy test within 7 days of study enrollment. Men and women with reproductive potential must use an effective contraceptive method while enrolled in this study and for 3 months after the patient has completed study.
* Patient must be able to swallow.
* Signed, written informed consent from patient or guardian.
* Estimated life expectancy of at least 12 weeks.

Exclusion Criteria:

* Known sensitivity to study drug or its analogs.
* Treatment with any investigational therapy within the preceding 4 weeks.
* Patients with hematological malignancies including leukemia, lymphoma, or multiple myeloma.
* Active and uncontrolled infection.
* Psychiatric disorders, alcohol or chemical abuse that would interfere with consent or follow-up.
* Uncontrolled congestive heart failure or angina.
* Pregnancy or lactation.
* Any other severe concurrent disease, which as judged by the investigator, would make the patient inappropriate for entry into this study.
* Patients with active gastrointestinal bleeding or ulceration, unhealed wounds or active thrombosis.
* Patients who are on anticoagulant therapy or taking aspirin, nonsteroidal anti-inflammatory drugs, unfractionated heparin, low molecular weight heparin, danaproid, thrombolytic agents, anti-platelet antibodies, glycoprotein IIb, IIIa antagonists, H2 blockers, or proton pump inhibitors.
* Brain or leptomeningeal metastases.
* Patients known to be HIV positive or who have an AIDS-related illness.
* Patients with a history of gastrointestinal bleeding from varices, arteriovenous malformations, Osler Weber Rendu syndrome, polyps, prior surgery, or gastric ulcerations. Patients who had bleeding not associated with a coagulopathy after surgery or gastric ulceration and who have no further bleeding or recurrence of their ulcers for more than one year are eligible for this study.
* Patients with a total accumulated doxorubicin or equivalent dose over 450 mg/m2.
* Patients with more than 1 risk factor, where a risk factor is defined as any one of the following (1-7):1. prior anthracyclines larger than 300 mg/m2 doxorubicin equivalent.2.mediastinum/left breast irradiation. 3.history of arterial hypertension (systolic blood pressure greater than 140 or diastolic blood pressure greater than 90, or receiving anti-hypertensive treatment).4. obesity (body mass index (BMI)[30]).5. diabetes mellitus (fasting plasma glucose level greater than 126 mg/dL American Diabetes Association (ADA) guidelines).6. smoking (any smoking in the month prior to study entry).7. hypercholesterolemia (greater than 240 mg/dL).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Start 2001-05; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
MTD of NM-3 is the dose at which less than or equal to 1 of 6 patients experiences a DLT

SECONDARY OUTCOMES:
Anti-tumor activity
VEGF and bFGF in urine, plasma and serum
Circulating endothelial cells

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- Boston, Massachusetts, United States

REFERENCES:
- See also: Related Info — http://www.genzyme.com